CLINICAL TRIAL: NCT00378430
Title: " Patients Attitude Towards Physicians and Health Screening Issues Among First Generation Asian-Indian Immigrants to United States".
Status: Terminated | Type: Observational
Why Stopped: poor response to questionnaire
Sponsor: University of California, San Francisco (Other)
Other Study IDs: 200654
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Health Screening

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Aim - To better understand expectations and attitudes of first generation immigrants from India to USA.

Background - The is large difference in healthcare system as practiced in India and in USA. Most people who have lived in India for certain period of their life have basic understanding of health-care system in India. In general it is the physician who makes choices for patients there , also the concept of health screening is less prevalent. After immigrating to USA these immigrants are exposed to new healthcare system. We donot have any data showing their attitudes to some specific questions and physician preference in general. We also have significant concentration of these ethnic group in the central valley.

With this questionnaire study we hope to get better understanding of their beliefs and expectations. We have tried to keep the questions simple and straightforward.

ELIGIBILITY:
Inclusion Criteria:

* First generation immigrants from India to USA
* Currently living in USA
* Planning to live in USA and utilize local healthcare facilities

Exclusion Criteria:

* Age < 18
* People born in USA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harminder Longia, MD, Study Director — University of California, San Francisco
Locations (1):
- UCSF , Fresno, Fresno, California, United States